CLINICAL TRIAL: NCT03805672
Title: Is Therapeutic Anticoagulation Necessary for the Treatment of Distal Deep Venous Thrombosis of the Lower Extremity? A Randomized, Controlled Trial
Brief Title: Below Knee DVT Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to low enrollment because of decrease in DVT rates.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Martin A Schreiber, MD, Professor & Chief of Trauma, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9134
Record Dates: First submitted 2015-01-14; First posted 2019-01-16 (Actual); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Deep Vein Thrombosis (DVT); Blood Clots
Keywords: Lovenox; enoxaparin; DVT
MeSH Terms: conditions — Venous Thrombosis; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose Enoxaparin (Active Comparator): Subjects are randomized to receive or begin prophylactic dosing (30 mg BID) of enoxaparin for 6 weeks or until DVT resolution.
  Interventions: Drug: Low Dose Enoxaparin
- High Dose Enoxaparin (Active Comparator): Subjects are randomized to begin therapeutic dosing (1 mg/kg body weight BID) of enoxaparin for 6 weeks or until DVT resolution.
  Interventions: Drug: High Dose Enoxaparin

INTERVENTIONS:
Drug: Low Dose Enoxaparin
  Other Names: Lovenox
  Arms: Low Dose Enoxaparin
Drug: High Dose Enoxaparin
  Other Names: Lovenox
  Arms: High Dose Enoxaparin

SUMMARY:
Hospitalized patients are at risk of developing blood clots in the legs (Deep Vein Thrombosis or DVT), which can lead to death if those clots break off and migrate to the lungs. We know that if there is a blood clot in the large leg veins near the hips and in the thighs, treating these patients with high-doses of blood thinners reduces the risk of these deaths.

It is unclear if treating blood clots in the calf with high doses of blood thinners is better than using low doses. In this study, after being diagnosed with a blood clot in the calf, patients will be treated with either low dose or high dose enoxaparin (Lovenox), a blood thinner. We will then see if low dose blood thinner has similar results as high dose blood thinner.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 admitted to a trauma or general surgery service will be eligible
* Patients diagnosed with an isolated distal DVT
* Able to obtain informed consent

Exclusion Criteria:

* Patients with a previous diagnosis of hypercoagulability
* Patients on chronic anticoagulation
* Patients with a history of heparin induced thrombocytopenia
* Patients have preexisting contraindications to anticoagulation
* Patients in renal failure requiring adjusted enoxaparin dosing
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schreiber, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18 years or older who were admitted to the trauma or other surgical service and diagnosed during their hospital admission with an isolated distal DVT were invited to participate in the study.
Groups:
- Low Dose Enoxaparin: Subjects are randomized to receive or begin prophylactic dosing (30 mg BID) of enoxaparin for 6 weeks or until DVT resolution.
  Low Dose Enoxaparin
- High Dose Enoxaparin: Subjects are randomized to begin therapeutic dosing (1 mg/kg body weight BID) of enoxaparin for 6 weeks or until DVT resolution.
  High Dose Enoxaparin
Period: Overall Study
Arm/Group | Low Dose Enoxaparin | High Dose Enoxaparin
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Enoxaparin | High Dose Enoxaparin | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (38.2) | 59.5 (37.5) | 52.3 (32.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Deep Vein Thrombosis Resolution
Description: Evaluation of DVT resolution
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Enoxaparin | High Dose Enoxaparin
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Low Dose Enoxaparin | High Dose Enoxaparin
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Enoxaparin (N=2) | High Dose Enoxaparin (N=2)
Bleeding at incision site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Subject experienced some increased bleeding at the incision site on lower extremity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No